CLINICAL TRIAL: NCT05013736
Title: Perinatal Stroke: Longitudinal Assessment of Infant Brain Organization and Recovery Through Neuroexcitability, Neuroimaging and Motor Development
Brief Title: Baby Brain Recovery Study
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2021-0412; A536761 (Other: UW Madison); SMPH/PEDIATRICS/PEDIATRICS (Other: UW Madison); Protocol ver 15 (Other: UW Madison); 7R01HD098202-02 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Perinatal Stroke
Keywords: Magnetic Resonance Imaging (MRI); Brain Reorganization; Brain Lesions; perinatal stroke; neonatal hemorrhagic stroke; neonatal thrombotic stroke; neonatal intracranial hemorrhage; neonatal periventricular leukomalacia; hypoxic ischemic encephalopathy; neonatal brain bleed; early brain injury
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Brain Injuries | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Infants: Pre-term and term born infants with corrected gestational age between term age and 24 months with radiologically-confirmed acute unilateral or bilateral brain lesions, including perinatal stroke, neonatal hemorrhagic or thrombotic stroke, involving the motor cortex and/or subcortical structures, and intracranial hemorrhage, involving the motor cortex and/or subcortical white matter, or periventricular leukomalacia. Parents/legal guardians able to attend study visits at the University of Wisconsin-Madison.
  Interventions: Device: Magnetic Resonance Imaging; Behavioral: Behavioral Assessments; Device: Non invasive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Magnetic Resonance Imaging — 3 Tesla Discovery MR750 MRI scanner (GE Healthcare, Waukesha, WI) will be used to perform structural imaging, diffusion MRI, relaxometry and microstructural imaging. The exact scan length and parameters of each scan type (T1, T2, DWI) will be set for this study to optimize the quality of data and decrease the length of scanning session for each type of scan. All of the imaging methods have been previously implemented at UW-Madison. Each sequence will take approximately 5-10 minutes.
  Other Names: MRI
Behavioral: Behavioral Assessments — The behavioral assessments (GMA: General Movements Assessment; HINE: Hammersmith Infant Neurological Examination; Baby Observation of Selective Control AppRaisal (BabyOSCAR); Bayley-4 / Bayley Scales of Infant and Toddler Development 4th ed; Pediatric Evaluation of Disability Inventory -Computer Adaptive Test (PEDI-CAT)) are infant and age-specific and will be administered by trained pediatric occupational and physical therapists.
Device: Non invasive Transcranial Magnetic Stimulation — TMS will be used to assess cortical excitability and circuitry (not as a neuromodulation intervention). Single-pulse TMS (Magstim 200², Magstim, UK) with a scalp surface coil will be used to assess how the brain is developing and how connected the tract is, between the brain and a target muscle on the arm. 10-20 TMS stimulation pulses will be delivered at a range of stimulation intensities (50-100%) increasing by 5% maximal stimulator output (MSO) at each stage. After this assessment, a brief assessment of peripheral nerve excitability will be performed. Peripheral stimulation will begin at 40% MSO. Stimulation intensity will be adjusted in increments of 5% until motor responses are evident on the EMG. Once motor responses are identified, 10 pulses will be delivered at the stimulation intensity that produced the response. In sum, around 150 stimulation pulses per hemisphere of brain stimulation and 22-60 pulses of peripheral stimulation are expected for TMS assessment of each infant.
  Other Names: TMS

SUMMARY:
This study will be a longitudinal multiple-visit observational study, done to identify possible bioindicators of recovery and repair of motor corticospinal pathways which may be targeted by future interventions in infants with perinatal stroke.

65 participants will be recruited and complete 1 visit at time point 1 (0-2 months), and 2 visits at each timepoints 2-5 with windows of +- 4 weeks (3-6 months, 12 months, 18 months and 24 months). Visits will consist of Magnetic Resonance Imaging (MRI) assessment during the child's natural sleep, Transcranial Magnetic Stimulation (TMS), and Motor Behavioral Assessments.

DETAILED DESCRIPTION:
Perinatal stroke has disabling consequences; 50-75% of individuals will develop life-long motor impairment, and 10-60% will also have cognitive deficits. These deficits lead to challenges in the school and home environments, with decreased likelihood of employment and independence and increased caregiver burden. Additionally, perinatal stroke is one of the primary causes of cerebral palsy (CP), a chronic and disabling neurological condition affecting motor function.

The first two years of life constitute a critical period of brain development and heightened neuroplasticity. There is now a consensus that, due to brain plasticity and rapid development, providing an early intervention may result in optimal recovery and lower costs of care. Unfortunately, researchers still have only limited understanding of how the brain develops after perinatal stroke and as a result CP diagnoses are typically not made until two years of age. There is an urgent need for very early diagnosis, prognosis and understanding of mechanisms in order to develop novel early interventions to improve outcomes in perinatal stroke with resultant CP.

Integrating study team's experience in studying and caring for this vulnerable infant stroke population, they propose to use non-invasive brain stimulation, neuroimaging, and behavioral assessments to analyze associations between development patterns, especially in the CST, and potential diagnosis of CP.

Specific aims of this study are:

* Aim 1. Map the presence and excitability of corticospinal pathways.
* Aim 2. Map the structural integrity and connectivity of corticospinal pathways.
* Aim 3. Compare motor outcomes from clinical behavioral assessments against corticospinal tract excitability and integrity.
* Aim 4. Identify the association between brain white-matter connectivity and general movements.
* Aim 5. Identify the association between corticospinal circuitry and general movements.

Protocol Amendment approved on 10/22/2021 removes TMS intervention and outcomes, adds a study time point at 0-2 months, and lowers the eligibility age to term.

Protocol Amendment approved on 12/21/2021 adds the TMS intervention back.

ELIGIBILITY:
Main Inclusion Criteria:

* Infants with corrected gestational age between term age and 24 months of age at study enrollment
* Radiologically-confirmed acute unilateral or bilateral brain lesions, including perinatal stroke, neonatal hemorrhagic or thrombotic stroke, involving the motor cortex and/or subcortical structures, and intracranial hemorrhage, involving the motor cortex and/or subcortical white matter, periventricular leukomalacia, and hypoxic-ischemic encephalopathy (HIE)
* English-speaking parent/legal guardian (able to provide consent)

Main Exclusion Criteria:

* Other neurologic disorders unrelated to perinatal stroke/brain bleed/HIE
* Metabolic disorders
* Disorders of Cellular Migration and Proliferation
* Acquired Traumatic Brain Injury

Ages: 0 Years to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pre-term and term born infants with corrected gestational age between term age and 24 months with radiologically-confirmed acute unilateral or bilateral brain lesions, including perinatal stroke, neonatal hemorrhagic or thrombotic stroke, involving the motor cortex and/or subcortical structures, and intracranial hemorrhage, involving the motor cortex and/or subcortical white matter, or periventricular leukomalacia. Parents/legal guardians and infants able to attend study visits at the University of Wisconsin-Madison.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Cortical excitability measured as presence/absence of motor evoked potentials (MEP) | 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
  Motor evoked potentials (MEPs) are the electrical signals recorded from the descending motor pathways or from muscles following stimulation of motor pathways within the brain.
  Responses from TMS pulses will be measured by recording muscle activity, referred to as motor evoked potentials (MEP).
Change in Cortical excitability measured by intensity of motor threshold (MT) | 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
  The MT is the minimum stimulation intensity that will elicit a consistent MEP of a pre-determined amplitude. MT and MEP are the common measures of TMS-induced excitability. Together, these measures provide information about the brain's excitability, associated with synaptic activity.
Change in Mean Fractional Anisotropy (FA) within the CST | 1 ±1 month, 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
  Mean Fractional Anisotropy (FA) within the CST will be used to study structural connectivity. It is a dimensionless index between 0 and 1. (0 equals no anisotropy; greater anisotropy is indicated by higher FA values approaching the maximum of 1).
  N=10 infants aged 0-2 months (first timepoint) will participate in MRI scans
Behavioral assessments: General Movements Assessment (GMA) reported on binary (Y/N) scale | 1 ±1 month
  The General Movements Assessment is used to identify absent or abnormal general movements. GMA requires 5-10 minutes video taping when infants are placed in spine position for scoring.
  "Absence or abnormal movements" will be reported as "Y".
Behavioral assessments: General Movements Assessment (GMA) reported on binary (Y/N) scale | 3 ±1 months
  The General Movements Assessment is used to identify absent or abnormal general movements. GMA requires 5-10 minutes video taping when infants are placed in spine position for scoring.
  "Absence or abnormal movements" will be reported as "Y".
Behavioral assessments: Hammersmith Infant Neurological Examination (HINE) global score | 1 ±1 month
  The HINE includes three sections, the Neurological Examination, the Development of Motor Functions and the State of Behaviour. The first section evaluates cranial nerve, posture, movements, tone and reflexes. These items are not age-dependent. The second section evaluates head control, sitting, voluntary grasping, rolling, crawling and walking. The third section evaluates state of consciousness, emotional state and social orientation.
  The maximum score for any one item is a score of 3 and the minimum is a score of 0. A subscore can be given for each section and the overall global score can be calculated by summing up all 26 items (range: 0-78), with higher scores indicating better neurological performance. High-risk cutoff scores for cerebral palsy are <57 at 3 months and <73 at 6, 9, or 12 months. See Novak et al, 2017 linked in the reference section for context.
Behavioral assessments: Hammersmith Infant Neurological Examination (HINE) global score | 3-6 months (one visit in this time frame)
  The HINE includes three sections, the Neurological Examination, the Development of Motor Functions and the State of Behaviour. The first section evaluates cranial nerve, posture, movements, tone and reflexes. These items are not age-dependent. The second section evaluates head control, sitting, voluntary grasping, rolling, crawling and walking. The third section evaluates state of consciousness, emotional state and social orientation.
  The maximum score for any one item is a score of 3 and the minimum is a score of 0. A subscore can be given for each section and the overall global score can be calculated by summing up all 26 items (range: 0-78), with higher scores indicating better neurological performance. High-risk cutoff scores for cerebral palsy are <57 at 3 months and <73 at 6, 9, or 12 months. See Novak et al, 2017 linked in the reference section for context.
Behavioral assessments: Hammersmith Infant Neurological Examination (HINE) global score | 12±1 months
  The HINE includes three sections, the Neurological Examination, the Development of Motor Functions and the State of Behaviour. The first section evaluates cranial nerve, posture, movements, tone and reflexes. These items are not age-dependent. The second section evaluates head control, sitting, voluntary grasping, rolling, crawling and walking. The third section evaluates state of consciousness, emotional state and social orientation.
  The maximum score for any one item is a score of 3 and the minimum is a score of 0. A subscore can be given for each section and the overall global score can be calculated by summing up all 26 items (range: 0-78), with higher scores indicating better neurological performance. High-risk cutoff scores for cerebral palsy are <57 at 3 months and <73 at 6, 9, or 12 months. See Novak et al, 2017 linked in the reference section for context.
Behavioral assessments: Hammersmith Infant Neurological Examination (HINE) global score | 18±1 months
  The HINE includes three sections, the Neurological Examination, the Development of Motor Functions and the State of Behaviour. The first section evaluates cranial nerve, posture, movements, tone and reflexes. These items are not age-dependent. The second section evaluates head control, sitting, voluntary grasping, rolling, crawling and walking. The third section evaluates state of consciousness, emotional state and social orientation.
  The maximum score for any one item is a score of 3 and the minimum is a score of 0. A subscore can be given for each section and the overall global score can be calculated by summing up all 26 items (range: 0-78), with higher scores indicating better neurological performance. High-risk cutoff scores for cerebral palsy are <57 at 3 months and <73 at 6, 9, or 12 months. See Novak et al, 2017 linked in the reference section for context.
Behavioral assessments: Hammersmith Infant Neurological Examination (HINE) global score | 24±1 months
  The HINE includes three sections, the Neurological Examination, the Development of Motor Functions and the State of Behaviour. The first section evaluates cranial nerve, posture, movements, tone and reflexes. These items are not age-dependent. The second section evaluates head control, sitting, voluntary grasping, rolling, crawling and walking. The third section evaluates state of consciousness, emotional state and social orientation.
  The maximum score for any one item is a score of 3 and the minimum is a score of 0. A subscore can be given for each section and the overall global score can be calculated by summing up all 26 items (range: 0-78), with higher scores indicating better neurological performance. High-risk cutoff scores for cerebral palsy are <57 at 3 months and <73 at 6, 9, or 12 months. See Novak et al, 2017 linked in the reference section for context.
Behavioral assessments: Hammersmith Infant Neurological Examination (HINE) Asymmetry Scores | data collected at 1 ±1 month, 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
  An asymmetry can also be recorded for each item, with one point maximum allotted per item, with a total score ranging from 0-26. Based on the literature regarding asymmetries, the cutoff score of >3 asymmetries will be used for recommendation of referral to early intervention service. See article by Fehlings, 2024 for additional context.
Behavioral assessments: Bayley Scales of Infant and Toddler Development Test, 4th edition (Bayley-4) score | 3-6 months (one visit in this time frame)
  Bayley-4 is a developmental test that measures cognitive, language, motor, and social-emotional domains of infants and young children between 1 and 42 months of age. A higher score generally corresponds with higher function.
Behavioral assessments: Bayley Scales of Infant and Toddler Development Test, 4th edition (Bayley-4) score | 12±1 months
  Bayley-4 is a developmental test that measures cognitive, language, motor, and social-emotional domains of infants and young children between 1 and 42 months of age. A higher score generally corresponds with higher function.
Behavioral assessments: Bayley Scales of Infant and Toddler Development Test, 4th edition (Bayley-IV) score | 18±1 months
  Bayley-4 is a developmental test that measures cognitive, language, motor, and social-emotional domains of infants and young children between 1 and 42 months of age. A higher score generally corresponds with higher function.
Behavioral assessments: Bayley Scales of Infant and Toddler Development Test, 4th edition (Bayley-4) score | 24±1 months
  Bayley-4 is a developmental test that measures cognitive, language, motor, and social-emotional domains of infants and young children between 1 and 42 months of age. A higher score generally corresponds with higher function.
Baby Observation of Selective Control AppRaisal (Baby OSCAR) | 1±1 month
  Baby OSCAR assessments are scored from video recordings of infant movement. Each limb is scored separately, with scores ranging 0-7 per lower limb, and 0-9 per upper limb for a total score of 0-32. Higher scores indicate better selective motor control.
Baby Observation of Selective Control AppRaisal (Baby OSCAR) | 3-6 months (one visit in this time frame)
  Baby OSCAR assessments are scored from video recordings of infant movement. Each limb is scored separately, with scores ranging 0-7 per lower limb, and 0-9 per upper limb for a total score of 0-32. Higher scores indicate better selective motor control.
Change in Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) | 1 ±1 month, 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
  Patient/caregiver-reported outcome measure of functional abilities and performance in children with disabilities. Scores are displayed instantly after completion of an assessment. A Detailed Score Report and a Summary Score Report are available. Normative scores are provided as age percentiles and T scores are based on a child's chronological age and intended for use by clinicians so that they may interpret a particular child's functioning relative to others of the same age. Scaled scores provide a way to look at a child's current functional skills and progress in these skills over time. Scaled scores are especially helpful in documenting improvements in functional skills for children not expected to exhibit or regain normative levels of functioning.

SECONDARY OUTCOMES:
Change in blood pressure | 1 ±1 month, 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
Change in heart rate | 1 ±1 month, 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
Change in skin integrity reported as presence/absence of skin redness/rash | 1 ±1 month, 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
Change in body temperature | 1 ±1 month, 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
Change in respiration rate | 1 ±1 month, 3-6 months (one visit in this time frame), 12±1 months, 18±1 months, 24±1 months
  Respiration rate will be measured as breaths/minute.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Gillick, PhD, MSPT, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial will be shared after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months after publication of primary outcomes, and ending 5 years after that date
Access Criteria: Data will be shared with the researchers whose proposed use of the data is for independent verification of study outcomes or to conduct subsequent clinical research. Data sharing will be approved by an independent review committee identified for this purpose.
  Proposals should be directed to bgillick@wisc.edu. If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

REFERENCES:
- [Background] Ganesan V, Hogan A, Shack N, Gordon A, Isaacs E, Kirkham FJ. Outcome after ischaemic stroke in childhood. Dev Med Child Neurol. 2000 Jul;42(7):455-61. doi: 10.1017/s0012162200000852. PMID 10972417
- [Background] Kirton A, Deveber G. Life after perinatal stroke. Stroke. 2013 Nov;44(11):3265-71. doi: 10.1161/STROKEAHA.113.000739. Epub 2013 Oct 8. No abstract available. PMID 24105698
- [Background] Herskind A, Greisen G, Nielsen JB. Early identification and intervention in cerebral palsy. Dev Med Child Neurol. 2015 Jan;57(1):29-36. doi: 10.1111/dmcn.12531. Epub 2014 Jul 9. PMID 25041565
- [Background] Novak I, Morgan C, Adde L, Blackman J, Boyd RN, Brunstrom-Hernandez J, Cioni G, Damiano D, Darrah J, Eliasson AC, de Vries LS, Einspieler C, Fahey M, Fehlings D, Ferriero DM, Fetters L, Fiori S, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Kakooza-Mwesige A, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Maitre N, McIntyre S, Noritz G, Pennington L, Romeo DM, Shepherd R, Spittle AJ, Thornton M, Valentine J, Walker K, White R, Badawi N. Early, Accurate Diagnosis and Early Intervention in Cerebral Palsy: Advances in Diagnosis and Treatment. JAMA Pediatr. 2017 Sep 1;171(9):897-907. doi: 10.1001/jamapediatrics.2017.1689. PMID 28715518
- [Background] Lemon RN. Descending pathways in motor control. Annu Rev Neurosci. 2008;31:195-218. doi: 10.1146/annurev.neuro.31.060407.125547. PMID 18558853
- [Background] Cioni G, D'Acunto G, Guzzetta A. Perinatal brain damage in children: neuroplasticity, early intervention, and molecular mechanisms of recovery. Prog Brain Res. 2011;189:139-54. doi: 10.1016/B978-0-444-53884-0.00022-1. PMID 21489387
- [Background] Frye RE, Rotenberg A, Ousley M, Pascual-Leone A. Transcranial magnetic stimulation in child neurology: current and future directions. J Child Neurol. 2008 Jan;23(1):79-96. doi: 10.1177/0883073807307972. Epub 2007 Dec 3. PMID 18056688
- [Background] Chen CY, Georgieff M, Elison J, Chen M, Stinear J, Mueller B, Rao R, Rudser K, Gillick B. Understanding Brain Reorganization in Infants With Perinatal Stroke Through Neuroexcitability and Neuroimaging. Pediatr Phys Ther. 2017 Apr;29(2):173-178. doi: 10.1097/PEP.0000000000000365. PMID 28350777
- [Background] Gillick BT, Gordon AM, Feyma T, Krach LE, Carmel J, Rich TL, Bleyenheuft Y, Friel K. Non-Invasive Brain Stimulation in Children With Unilateral Cerebral Palsy: A Protocol and Risk Mitigation Guide. Front Pediatr. 2018 Mar 16;6:56. doi: 10.3389/fped.2018.00056. eCollection 2018. PMID 29616203
- [Background] Nemanich ST, Chen CY, Chen M, Zorn E, Mueller B, Peyton C, Elison JT, Stinear J, Rao R, Georgieff M, Menk J, Rudser K, Gillick B. Safety and Feasibility of Transcranial Magnetic Stimulation as an Exploratory Assessment of Corticospinal Connectivity in Infants After Perinatal Brain Injury: An Observational Study. Phys Ther. 2019 Jun 1;99(6):689-700. doi: 10.1093/ptj/pzz028. PMID 30806664
- [Background] Allen CH, Kluger BM, Buard I. Safety of Transcranial Magnetic Stimulation in Children: A Systematic Review of the Literature. Pediatr Neurol. 2017 Mar;68:3-17. doi: 10.1016/j.pediatrneurol.2016.12.009. Epub 2017 Jan 4. PMID 28216033
- [Background] Chen CY, Rich TL, Cassidy JM, Gillick BT. Corticospinal Excitability in Children with Congenital Hemiparesis. Brain Sci. 2016 Oct 20;6(4):49. doi: 10.3390/brainsci6040049. PMID 27775599
- [Background] Roze E, Harris PA, Ball G, Elorza LZ, Braga RM, Allsop JM, Merchant N, Porter E, Arichi T, Edwards AD, Rutherford MA, Cowan FM, Counsell SJ. Tractography of the corticospinal tracts in infants with focal perinatal injury: comparison with normal controls and to motor development. Neuroradiology. 2012 May;54(5):507-16. doi: 10.1007/s00234-011-0969-5. Epub 2011 Oct 18. PMID 22006424
- [Background] van der Aa NE, Northington FJ, Stone BS, Groenendaal F, Benders MJ, Porro G, Yoshida S, Mori S, de Vries LS, Zhang J. Quantification of white matter injury following neonatal stroke with serial DTI. Pediatr Res. 2013 Jun;73(6):756-62. doi: 10.1038/pr.2013.45. Epub 2013 Mar 11. PMID 23478641
- [Background] Adde L, Rygg M, Lossius K, Oberg GK, Stoen R. General movement assessment: predicting cerebral palsy in clinical practise. Early Hum Dev. 2007 Jan;83(1):13-8. doi: 10.1016/j.earlhumdev.2006.03.005. Epub 2006 May 2. PMID 16650949
- [Background] Yu YT, Hsieh WS, Hsu CH, Chen LC, Lee WT, Chiu NC, Wu YC, Jeng SF. A psychometric study of the Bayley Scales of Infant and Toddler Development - 3rd Edition for term and preterm Taiwanese infants. Res Dev Disabil. 2013 Nov;34(11):3875-83. doi: 10.1016/j.ridd.2013.07.006. Epub 2013 Sep 9. PMID 24029804
- [Background] Peyton C, Yang E, Msall ME, Adde L, Stoen R, Fjortoft T, Bos AF, Einspieler C, Zhou Y, Schreiber MD, Marks JD, Drobyshevsky A. White Matter Injury and General Movements in High-Risk Preterm Infants. AJNR Am J Neuroradiol. 2017 Jan;38(1):162-169. doi: 10.3174/ajnr.A4955. Epub 2016 Oct 27. PMID 27789448
- [Background] Romeo DM, Ricci D, Brogna C, Mercuri E. Use of the Hammersmith Infant Neurological Examination in infants with cerebral palsy: a critical review of the literature. Dev Med Child Neurol. 2016 Mar;58(3):240-5. doi: 10.1111/dmcn.12876. Epub 2015 Aug 25. PMID 26306473
- [Background] Chen CY, Tafone S, Lo W, Heathcock JC. Perinatal stroke causes abnormal trajectory and laterality in reaching during early infancy. Res Dev Disabil. 2015 Mar;38:301-8. doi: 10.1016/j.ridd.2014.11.014. Epub 2015 Jan 9. PMID 25577180
- [Background] Dean DC 3rd, Dirks H, O'Muircheartaigh J, Walker L, Jerskey BA, Lehman K, Han M, Waskiewicz N, Deoni SC. Pediatric neuroimaging using magnetic resonance imaging during non-sedated sleep. Pediatr Radiol. 2014 Jan;44(1):64-72. doi: 10.1007/s00247-013-2752-8. Epub 2013 Aug 6. PMID 23917588
- [Background] Kowalski JL, Nemanich ST, Nawshin T, Chen M, Peyton C, Zorn E, Hickey M, Rao R, Georgieff M, Rudser K, Gillick BT. Motor Evoked Potentials as Potential Biomarkers of Early Atypical Corticospinal Tract Development in Infants with Perinatal Stroke. J Clin Med. 2019 Aug 13;8(8):1208. doi: 10.3390/jcm8081208. PMID 31412592
- [Background] Fehlings D, Makino A, Church P, Banihani R, Thomas K, Luther M, Lam-Damji S, Vollmer B, Haataja L, Cowan F, Romeo DM, George J, Kumar S. The Hammersmith Infant Neurological Exam Scoring Aid supports early detection for infants with high probability of cerebral palsy. Dev Med Child Neurol. 2024 Sep;66(9):1255-1257. doi: 10.1111/dmcn.15977. Epub 2024 May 31. No abstract available. PMID 38818710
- [Derived] Casey CP, Sutter EN, Grimaldo A, Collins KM, Guerrero-Gonzalez J, McAdams RM, Dean DC 3rd, Gillick BT. Preservation of Bilateral Corticospinal Projections from Injured Hemisphere After Perinatal Stroke. Brain Sci. 2025 Jan 17;15(1):82. doi: 10.3390/brainsci15010082. PMID 39851449
- See also: Link to ClinicalTrials.gov record of the pilot study which lead to current study — https://clinicaltrials.gov/ct2/show/NCT02743728?term=Transcranial+Magnetic+Stimulation&recrs=ab&cond=Perinatal+Stroke&draw=2&rank=1